CLINICAL TRIAL: NCT06241274
Title: Clinical Study of Moxibustion in the Treatment of Hemorrhagic Cystitis After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Moxibustion in the Treatment of Hemorrhagic Cystitis After Allo-HSCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yi Zhang, physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT230698
Record Dates: First submitted 2024-01-07; First posted 2024-02-05 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Moxibustion; Hematopoietic Stem Cell Transplantation; Hemorrhagic Cystitis; Treatment
MeSH Terms: conditions — Cystitis, Hemorrhagic | interventions — Moxibustion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moxibustion (Experimental): Subjects received symptomatic supportive treatment combined with moxibustion covering Shenque, Zhonggong, Guanyuan, and Qihai for 30 minutes every day for 14 days.
  Interventions: Other: Moxibustion; Other: Symptomatic supportive treatment

INTERVENTIONS:
Other: Moxibustion — Subjects received moxibustion covering Shenque, Zhonggong, Guanyuan, and Qihai for 30 minutes every day for 14 days.
Other: Symptomatic supportive treatment — Symptomatic supportive treatment.

SUMMARY:
This study was a prospective, multicenter, single-arm clinical study planned to enroll 60 patients who developed hemorrhagic cystitis after sexually allogeneic hematopoietic stem cell transplantation Patients with hemorrhagic cystitis after allogeneic hematopoietic stem cell transplantation were given symptomatic supportive treatment combined with moxibustion covering Shenque, Zhongguo, Guanyuan, and Qihai for 30 minutes every day for 14 days and urine routine was collected every day for 14 days to assess the severity of hemorrhagic cystitis and pain scores to evaluate the effectiveness of moxibustion in treating hemorrhagic cystitis after allogeneic hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. patients were fully aware of the study, participated voluntarily, and signed the informed consent form;
2. Age: 18-55 years old;
3. patients with hemorrhagic cystitis after allogeneic hematopoietic stem cell transplantation;

Exclusion Criteria:

1. refusal to participate in this clinical study;
2. broken or sensitized skin corresponding to the moxibustion site;
3. allogeneic hematopoietic stem cell transplantationpatients pretreated with the Reduced-intensity conditioning.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Core Lower Urinary Tract Symptom Score | 14 days
  The Core Lower Urinary Tract Symptom Score consists of 10 questions. Frequent daytime urination---0 points:<7 times;1 point:8~9 times;2 points:10~14 times;3 points:> 14 times. Nocturia---0 points:0 times/night;1 point:1 time/night;2 points: 2~3 times/night;3 points:> 3 times/night. The other 8 problems were urgency, dysuria, hesitancy, thin urine line, urge incontinence, stress incontinence, bladder pain, and urethral pain, which were rated as 0, 1, 2, and 3 according to their frequency (never, rarely, sometimes, and often).

CONTACTS AND LOCATIONS:
Locations (1):
- Yi Zhang, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang AK, Foca MD, Jin Z, Vasudev R, Laird M, Schwartz S, Qureshi M, Kolb M, Levinson A, Bhatia M, Kung A, Garvin J, George D, Della-Latta P, Whittier S, Saiman L, Satwani P. Bacterial bloodstream infections in pediatric allogeneic hematopoietic stem cell recipients before and after implementation of a central line-associated bloodstream infection protocol: A single-center experience. Am J Infect Control. 2016 Dec 1;44(12):1650-1655. doi: 10.1016/j.ajic.2016.04.229. Epub 2016 Jul 1. PMID 27378008
- [Background] Mackall C, Fry T, Gress R, Peggs K, Storek J, Toubert A; Center for International Blood and Marrow Transplant Research (CIBMTR); National Marrow Donor Program (NMDP); European Blood and Marrow Transplant Group (EBMT); American Society of Blood and Marrow Transplantation (ASBMT); Canadian Blood and Marrow Transplant Group (CBMTG); Infectious Disease Society of America (IDSA); Society for Healthcare Epidemiology of America (SHEA); Association of Medical Microbiology and Infectious Diseases Canada (AMMI); Centers for Disease Control and Prevention (CDC). Background to hematopoietic cell transplantation, including post transplant immune recovery. Bone Marrow Transplant. 2009 Oct;44(8):457-62. doi: 10.1038/bmt.2009.255. No abstract available. PMID 19861978
- [Background] Gutierrez-Aguirre CH, Esparza-Sandoval AC, Palomares-Leal A, Jaime-Perez JC, Gomez-Almaguer D, Cantu-Rodriguez OG. Outpatient haploidentical hematopoietic stem cell transplant using post-transplant cyclophosphamide and incidence of hemorrhagic cystitis. Hematol Transfus Cell Ther. 2022 Apr-Jun;44(2):163-168. doi: 10.1016/j.htct.2020.09.149. Epub 2020 Dec 4. PMID 33814347
- [Background] Dalianis T, Ljungman P. Full myeloablative conditioning and an unrelated HLA mismatched donor increase the risk for BK virus-positive hemorrhagic cystitis in allogeneic hematopoetic stem cell transplanted patients. Anticancer Res. 2011 Mar;31(3):939-44. PMID 21498717
- [Background] Hassan Z, Remberger M, Svenberg P, Elbander M, Omazic B, Mattsson J, Conrad R, Svahn BM, Ahlgren A, Sairafi D, Aschan J, Le Blanc K, Barkholt L, Ringden O. Hemorrhagic cystitis: a retrospective single-center survey. Clin Transplant. 2007 Sep-Oct;21(5):659-67. doi: 10.1111/j.1399-0012.2007.00705.x. PMID 17845642
- [Background] Arango M, Cardona D. Hemorrhagic Cystitis after Haploidentical Transplantation with Post-Transplantation Cyclophosphamide: Protective Effect of MESNA Continuous Infusion. Biol Blood Marrow Transplant. 2020 Aug;26(8):1492-1496. doi: 10.1016/j.bbmt.2020.04.028. Epub 2020 May 15. PMID 32417488
- [Background] Tang B, Zhang J, Yang Z, Lu Y, Xu Q, Chen X, Lin J. Moxibustion for Diarrhea-Predominant Irritable Bowel Syndrome: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Evid Based Complement Alternat Med. 2016;2016:5105108. doi: 10.1155/2016/5105108. Epub 2016 May 16. PMID 27293460
- [Background] Sun ZR, Wang CB, Yin HN, Luan YX, Liu YX, Gong RQ, Gong N, Wang BL, Miao CX. [Network Meta-analysis of acupuncture and moxibustion for allergic rhinitis]. Zhongguo Zhen Jiu. 2021 Nov 12;41(11):1295-302. doi: 10.13703/j.0255-2930.20200916-0002. Chinese. PMID 34762387
- [Background] Li X, Li ZM, Tan JY, Wang T, Chen JX, Chen X, Yang L, Suen LKP. Moxibustion for post-stroke urinary incontinence in adults: A systematic review and meta-analysis of randomized controlled trials. Complement Ther Clin Pract. 2021 Feb;42:101294. doi: 10.1016/j.ctcp.2020.101294. Epub 2020 Dec 24. PMID 33360387